CLINICAL TRIAL: NCT03368703
Title: Physiopathology of Lower Cortical Activation in COPD Patients: Contribution of Cortical Neuromodulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 5 Santé (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 5S_EXCCOM
Record Dates: First submitted 2016-12-19; First posted 2017-12-11 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Physiology
Keywords: COPD; Transcranial direct-current stimulation; Transcranial magnetic stimulation; Motor-evoked potentials; Inhibition; Muscle weakness
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Inhibition, Psychological; Muscle Weakness | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COPD patients (Experimental): COPD patients group
  Interventions: Device: Anodal transcranial direct-current-stimulation; Device: Sham transcranial direct-current-stimulation
- Healthy subjects (Active Comparator): Healthy subject group, matched with COPD patients group on age, weight and BMI
  Interventions: Device: Anodal transcranial direct-current-stimulation; Device: Sham transcranial direct-current-stimulation

INTERVENTIONS:
Device: Anodal transcranial direct-current-stimulation — 2mA / 20min Anodal and Sham tDCS over dominant M1. Anodal tDCS consists of 30s of ramp up followed by 20min of stimulation and 30s of ramp down.
Device: Sham transcranial direct-current-stimulation — Sham tDCS consists of only 30s of ramp up followed by 30s of ramp down and no further stimulation.
  Participants therefore have the same feeling for both modalities : slight itching due to the induced current at the beginning of the protocol (during around 30s) allowing no differentiation by the participant between the anodal or sham sessions.

SUMMARY:
Patients with COPD have lower cortical activation and higher cortical inhibitory levels. The purpose of this study is to test the reversibility the lower cortical activation by counterbalancing the increased cortical inhibitory levels with neuro-modulation.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) patients exhibit not only respiratory symptoms but also a peripheral muscular weakness. This weakness is characterized by a loss in strength, harmful for the patients' life quality and vital prognostic. Even if many papers have enlightened damages at a peripheral level, the muscular atrophy itself cannot totally explain the loss in force. Furthermore, the contractile properties of COPD muscles fibres are preserved. Consequently, it seems that the peripheral muscle weakness cannot only be explained by peripheral factors and central structures may be involved.

A recent work showed that during quadriceps voluntary contraction, cortical activation in COPD patients was significantly lower than in healthy subjects, contributing in the loss in strength. However, the pathophysiology underlying this loss of strength is still unclear and two hypotheses can be advanced: 1) the influence of anatomical lesions in the brain of COPD patients and 2) the particular metabolism of this population. Indeed, COPD patients show a reduced oxidative activity and an increased glycolytic contribution (decreased type I fibres and increased type II fibres, increased glycolytic enzymes activity, increased metabolites production). This specific metabolic may lead to an over-activation of type III-IV afferents, projecting onto somatosensory cortex sensitive to metabolites at a peripheral level, and produce inhibitory activity on the primary motor cortex, seat of the motor control. What is reported in the literature so far, is that COPD patients display increased cortical inhibitory values than healthy subjects.

Therefore, beyond understanding better the nervous mechanisms involved in the COPD's peripheral muscle weakness, the aim of this study is to counterbalance this increased cortical inhibitory level.

We hypothesize that modulating inhibitory processes at a cortical level would induced a reduction of inhibitions in patients with COPD and an increase in the force produced. In case this hypothesis would be verified, we will be able to confirm that this increased cortical level in COPD patients is reversible and may be a target for rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Health insurance
* Patients : COPD Gold II-IV
* Patients : No rehabilitation since at least 1 yrs
* Control : sedentary (< 9 Voorips)

Exclusion Criteria:

* Pregnant women
* Seizures
* Unable to give written consent
* Metalic object above shoulders
* Dermatological issue concerning surface electrodes
* Drugs influencing central nervous system
* Caffeine consumption > 4 coffee / day
* Neurological disorders
* Patients : recent exacerbation (< 4 weeks)

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Change in motor-evoked potentials | Baseline (pre-intervention) ; Post-Stim (immediately post-intervention) ; Post-30 (30min post-intervention)
  Cortical excitability

SECONDARY OUTCOMES:
Change in short-interval intracortical inhibition | Baseline (pre-intervention) ; Post-Stim (immediately post-intervention) ; Post-30 (30min post-intervention)
  Cortical inhibition level
Change in cortical silent period | Baseline (pre-intervention) ; Post-Stim (immediately post-intervention) ; Post-30 (30min post-intervention)
  Cortical inhibition level
Change in cortical voluntary activation | Baseline (pre-intervention) ; Post-Stim (immediately post-intervention) ; Post-30 (30min post-intervention)
  Motor command
Change in strength | Baseline (pre-intervention) ; Post-Stim (immediately post-intervention) ; Post-30 (30min post-intervention)
  Functional output

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Guerin, MD, Principal Investigator — 5 Santé
Locations (1):
- Cliniques du Souffle, Lodève, Herault, France

IPD SHARING:
Plan to Share IPD: No